CLINICAL TRIAL: NCT00402870
Title: Postoperative Analgesic Requirements for the ProSeal Laryngeal Mask Airway Versus the Tracheal Tube in Females Undergoing Gynecological Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Medical University Innsbruck, Christian Keller, MD, M.Sc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006-95
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2007-12

CONDITIONS: Intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Device: ProSeal LMA — ProSeal LMA vs Tracheal Tube
Device: ProSeal LMA, Tracheal Tube — ProSeal LMA vs Tracheal Tube

SUMMARY:
The ProSeal laryngeal mask airway is a relatively new airway device with a modified cuff to increase the seal and a drain tube to provide a channel for regurgitated fluid, prevention of gastric insufflation and insertion of a gastric tube. In the following randomized prospective double-blind trial, we test the hypothesis that the postoperative analgesic requirements is higher for the ProSeal laryngeal mask airway than the tracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* Female
* ASA I-II
* Age 18-75
* Elective laparoscopic surgery

Exclusion Criteria:

* Known or predicted difficult airway
* Oropharyngeal pathology
* Mouth opening < 3.0 cm
* A body mass index > 35 kg m-2
* Increased risk of aspiration
* Inability to communicate or understand the visual analogue scale
* Analgesics within 24 hours of surgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keller, MD, M.Sc., Principal Investigator — Dept of Anesthesia, Medical University Innsbruck
Locations (1):
- Dept of Anesthesia, Innsbruck, Innsbruck, Austria